CLINICAL TRIAL: NCT06440928
Title: Investigation of the Effect of Cervical Segmental Mobilization on Pain, Functionality, Grip Strength and Quality of Life in Patients With Chronic Lateral Epicondylitis
Brief Title: Results of Cervical Segmental Mobilization in Patients With Chronic Lateral Epicondylitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Halic University (Other)
Responsible Party: Principal Investigator, Mustafa Yığılıtaş, lecturer, Halic University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023/106
Record Dates: First submitted 2024-05-05; First posted 2024-06-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: Epicondylitis of the Elbow; Servical Segmental Mobilization
Keywords: Lateral epicondylitis; Servical segmental mobilization; Pain; Quality of life; Grip strenght; Functionality
MeSH Terms: conditions — Tennis Elbow; Pain

STUDY DESIGN:
Intervention Model Description: randomised controlled and experimental study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- intervention grup: standart treatment and segmental mobilization grup (Experimental): Mobilisation specifically on the C7 segment will be performed by the physiotherapist 2 times a week for 3 weeks, making decisions on the choice of key parameters including treatment technique, spinal level, degree, direction, side and duration.
  Interventions: Behavioral: mobilization; Other: standard treatment
- intervention grup : standart treatment and deep friction (Experimental): The patients were asked to stretch for 20 s with the other hand with the shoulder in internal rotation, elbow in extension, forearm in pronation, wrist in flexion and ulnar deviation. In the first week, stretching exercises were recommended to be performed 3 sets a day, 5⨯20 s in one set and 45 s rest interval before strengthening exercises. The application will be performed with the thumb in the transverse direction, with the pressure tolerated by the individual, for 10 minutes after numbness is obtained, the treatment lasts approximately 10-15 minutes.
  Interventions: Other: standard treatment; Other: deep friction
- intervention grup: standart treatment. (Experimental): The patients were asked to stretch for 20 s with the other hand with the shoulder in internal rotation, elbow in extension, forearm in pronation, wrist in flexion and ulnar deviation. In the first week, stretching exercises were recommended to be performed 3 sets a day, 5⨯20 s in one set and 45 s rest interval before strengthening exercises. Starting from the 2nd week of treatment, it will be requested to be performed 3 sets a day, 5⨯20 s in one set, 5⨯20 s before exercise and 5⨯20 s after exercise.
  Interventions: Other: standard treatment

INTERVENTIONS:
Behavioral: mobilization — mobilization and exercise to be applied to patients with chronic lateral epicondylitis
  Other Names: excersize
  Arms: intervention grup: standart treatment and segmental mobilization grup
Other: standard treatment — standard treatment
Other: deep friction — deep friction
  Arms: intervention grup : standart treatment and deep friction

SUMMARY:
The aim of our study was to investigate the effect of cervical segmental mobilization on pain, functionality, grip strength and quality of life in patients with chronic lateral epicondylitis. It was planned as a randomized controlled experimental study.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 25-44
* Being diagnosed with LE by a physician
* Not having any defined pathology in the cervical region
* No neurological problems in the upper extremities
* No history of cervical surgery

Exclusion Criteria:

* Those with a history of infection, tumor, trauma in the cervical area
* Fibromyalgia patients
* Congenital or acquired deformities of the upper extremity
* History of shoulder or elbow surgery or dislocation
* Cervical radiculopathy
* Having had Wiplash

Ages: 25 Years to 44 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2024-08-15 (Estimated); Study Completion 2024-10-15 (Estimated)

PRIMARY OUTCOMES:
Assessment of Pain | 3 weeks
  In the assessment of pain, the "Visuel Analog Scale (VAS)" will be used and people will be asked to indicate the severity of their pain in the last 24 hours on a 10 cm chart. Before and after the session, VAS will be evaluated and recorded with the values measured with algometer. According to the pain scale in VAS application; "0" means no pain and "10" means the presence of unbearable pain, while patients will be asked to mark the pain they feel numerically between 0-10.
Quality of Life Short Form-36 | 3 weeks
  The scale consists of 36 statements. The scale has 8 dimensions including physical functioning (FF), social functioning (SF), role limitations related to physical functioning (RRF), role limitations related to emotional problems (ERR), mental health (MS), vitality (C), bodily pain (BA) and general health perception (GS). Quality of life increases as the scores on the scale increase. Minimum score is 0 and maximum score is 100.
Assessment of Functionality | 3 weeks
  Duruöz Hand Index (DEI) specifically for rheumatoid arthritis patients. The index includes hand dexterity in the kitchen, during dressing, while maintaining personal hygiene, at work and other general movements. Participants rate 18 items from 0 (no difficulty) to 5 (impossible to do). The total score ranges from 0-90. A high score indicates impaired hand function.
Grip Strength | 3 weeks
  Grip strength will be evaluated with Jamar Hand Dynamometer. In the grip strength evaluations of the hand, measurements will be taken from both the patient and the healthy side. In the measurements made from the patient side, painless grip strength and maximum grip strength will be evaluated separately in the elbow flexion position and elbow extension position. On the healthy side, maximum grip strength will be evaluated in both positions. Patients will be positioned and evaluated according to the holding and gripping force of the dynamometer to be used. The patient will be asked to squeeze the dynamometer as strongly as possible for 5 seconds, first with the intact and then with the affected side, and 3 measurements will be made with one-minute breaks between the measurements and the averages will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Yalova University, Yalova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No